CLINICAL TRIAL: NCT02351024
Title: Study to Assess the Comparative Bioavailability and Pharmacokinetics of Naproxen From OXP005 Tablets (Test) And Naprosyn® Tablets (Reference) in Normal, Healthy, Adult Subjects
Brief Title: Phase I Study PK Study With OXP005 and Naprosyn
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Pharmascience Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: OXP005-001
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OXP005 (Experimental)
  Interventions: Drug: OXP005
- Naproxen (Active Comparator)
  Interventions: Drug: Naprosyn®

INTERVENTIONS:
Drug: OXP005
  Other Names: Naproxen
  Arms: OXP005
Drug: Naprosyn®
  Other Names: Naproxen
  Arms: Naproxen

SUMMARY:
The Sponsor is developing a new form of naproxen (the study drug, OXP005), for the potential treatment of rheumatic and painful conditions. The study will compare the study drug to an already marketed formulation of prescription strength naproxen (Naprosyn® the reference product) by looking at how a single dose of the drug is taken up by the body. The safety and tolerability of the drug will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and non-pregnant, non breast feeding healthy female subjects aged 18 to 55 years
* Body mass index 18.0 to 30.0 kg/m2

Exclusion Criteria:

* History of or current significant diseases or conditions including any disease or condition affecting the haematopoietic, cardiovascular, renal, hepatic, endocrine, pulmonary, central nervous, immunological, dermatological, gastrointestinal or any other body system

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparative bioavailability of naproxen as measured by Tmax, Cmax, AUC, half-life | Day 1 & Day 8 single dose crossover

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom